CLINICAL TRIAL: NCT04588519
Title: Transcutaneous Auricular Neurostimulation (tAN) to Mitigate Withdrawal Behaviors in Neonates With Opioid Withdrawal
Brief Title: tAN to Mitigate Withdrawal Behaviors in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090960; 1R43DA050360-01 (NIH)
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active Transcutaneous Auricular Neurostimulation (Experimental): Transcutaneous Auricular Neurostimulation programmed to a pulse width of 250ms; channel 1: 5 Hz, mean intensity 0.3±0.2 mA; channel 2: 100 Hz, mean intensity 0.6±0.2 mA
  Interventions: Device: Spark Biomedical Roo Transcutaneous Auricular Neurostimulation (tAN) System

INTERVENTIONS:
Device: Spark Biomedical Roo Transcutaneous Auricular Neurostimulation (tAN) System — Spark Roo tAN System programmed to a pulse width of 250ms; channel 1: 5 Hz, mean intensity 0.3±0.2 mA; channel 2: 100 Hz, mean intensity 0.6±0.2 mA.

SUMMARY:
This first in-human-neonates, open-label pilot trial is designed to determine whether use of tAN in newborns with NOWS receiving oral morphine allows for faster weaning of morphine and decrease morphine use altogether. Reducing Neonatal Opioid Withdrawal Syndrome (NOWS) symptoms may also help lessen or eliminate the need for opioid medication and shorten the length of the hospital stay. The neurostimulation device, currently called the Roo is a safe form of neurostimulation that uses sticker-like patches worn in and around the ear during the withdrawal period. The patches deliver a small and painless current of electrical pulses to the skin and underlying cranial nerves.

DETAILED DESCRIPTION:
This first in-human-neonates, open-label pilot trial is designed to determine whether use of tAN in newborns with NOWS receiving oral morphine allows for faster weaning of morphine and decrease morphine use altogether. After obtaining parental consent, tAN is delivered to the left ear in NOWS newborns who are on a stable morphine dose for >12h (control dose), using a disposable, multi-channel (Channel1: auricular branch of the vagus nerve (ABVN); Channel2: ATN) earpiece electrode (Spark Biomedical, Inc). 30-minutes of tAN is delivered one hour prior to scheduled morphine dose, up to four times daily for up to 12 days. The device is programmed to a pulse width of 250ms; channel 1: 5 Hz, mean intensity 0.3±0.2 milliamps (mA); channel 2: 100 Hz, mean intensity 0.6±0.2 mA. Nurses score the Finnegan Neonatal Abstinence Scoring Tool (FNAST) every 3h after feeding and morphine is weaned every 12h if FNAST scores <8.

ELIGIBILITY:
Inclusion Criteria:

* Neonates or infants with opioid withdrawal or Neonatal Abstinence Syndrome (NAS) who have withdrawal scores requiring morphine replacement therapy. They must be clinically stable, on minimal respiratory support (Continuous positive airway pressure (CPAP), nasal cannula, or room air), >33 weeks gestational age at enrollment, and currently receiving replacement therapy for opioid dependence.
* Stable neonates who are dependent on opioids, such as after extracorporeal membrane oxygenation, severe illness or brain injury, will be included in this study, as these neonates represent a population in which tAN could minimize withdrawal while not adding to burden of pharmacotherapies. Congenital syndromes may be included if the infants do not have major, unrepaired anomalies.

Exclusion Criteria:

1. Unstable infants or those requiring significant respiratory support.
2. Repeated episodes of autonomic instability (apnea or bradycardia) which are not self-resolving *
3. Infants <33weeks gestation at enrollment.
4. Major unrepaired congenital anomalies
5. Cardiomyopathy *Preterm infants commonly have short periods of shallow or absent breathing or lower heart rate termed apnea and bradycardia, respectively, and most are being treated for these physiologic manifestations of prematurity with caffeine, an effective central stimulant. Infants are on cardiorespiratory monitors through the nursery stay with recording devices to capture events and play them back. However, nearly all of these events are self resolving, meaning the infant resolves the breathing pause or bradycardia on their own. Infants who require repeated episodes of stimulation to come out of these events are defined as unstable. Similarly, infants on significant respiratory support are not stable, and will not be eligible.

Ages: 33 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share participant data

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Transcutaneous Auricular Neurostimulation: tAN therapy was administered for 30 minutes one hour prior to morphine administration, up to four times per day, for up to 12 days (or discontinuation of morphine; whichever came first).
  The Spark Roo tAN System was programmed to a pulse width of 250ms; channel 1: 5 Hz, mean intensity 0.3±0.2 mA; channel 2: 100 Hz, mean intensity 0.6±0.2 mA.
Period: Overall Study
Arm/Group | Active Transcutaneous Auricular Neurostimulation
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Transcutaneous Auricular Neurostimulation
Number analyzed (Participants) | 8
Age, Customized [Median (Full Range); unit: weeks]
  Gestational Age at Enrollment | 38.2 [35.1 to 43.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With no Adverse Events Related to Bradycardia (HR < 80 Bpm), Worsening of Swallowing or Feeding, Skin Irritation, or Elevation of Neonatal Infant Pain Scores.
Description: No adverse events of bradycardia (HR < 80 bpm), worsening of swallowing or feeding, skin irritation, or elevation of Neonatal Infant Pain Scores.
Time Frame: 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active Transcutaneous Auricular Neurostimulation
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Mean Finnegan Scores During Days of tAN Sessions
Description: The Finnegan Scale assesses 31 of the most common signs of neonatal drug withdrawal syndrome and is scored on the basis of pathological significance and severity of the adverse symptoms. Scores for each sign are added to obtain a total score. Total scores range from 0-20, where lower scores are indicative of less severe signs of neonatal drug withdrawal symptoms.
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcutaneous Auricular Neurostimulation
Number analyzed (Participants) | 8
score on a scale | 6.33 (0.98)

3. Secondary Outcome: Duration of Morphine Weaning
Description: Defined as the number of days between tAN therapy initiation and morphine discontinuation. A shorter duration of morphine weaning indicates better treatment efficacy.
Time Frame: 12 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Active Transcutaneous Auricular Neurostimulation
Number analyzed (Participants) | 8
Days | 6.0 [4.8 to 8.0]

4. Secondary Outcome: Length of Hospital Stay
Description: Defined as the number of days between birth and discharge. A shorter length of stay indicates better treatment efficacy.
Time Frame: From participant birth to hospital discharge, a median of 17 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Active Transcutaneous Auricular Neurostimulation
Number analyzed (Participants) | 8
Days | 17.0 [15.3 to 28.5]

ADVERSE EVENTS:
Time Frame: Through study completion (up to 12 days per participant)
Arm/Group | Active Transcutaneous Auricular Neurostimulation
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Transcutaneous Auricular Neurostimulation (N=8)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
This trial was open-label with no sham control group, limiting interpretation of the study results in terms of the placebo effect and true effect. An RCT would further address additional study limitations, namely the small sample size and conduct and a single center. The inclusion of infants at different durations of morphine therapy does not allow for interpretation of the potential effect of tAN during early administration of morphine therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT04588519/Prot_000.pdf